CLINICAL TRIAL: NCT02321293
Title: A Phase 1 Open-label Prospective Cohort Trial of Curcumin Plus Tyrosine Kinase Inhibitors for Epidermal Growth Factor Receptor (EGFR)-Mutant Advanced Non-small Cell Lung Cancer
Brief Title: A Open-label Prospective Cohort Trial of Curcumin Plus Tyrosine Kinase Inhibitors (TKI) for EGFR -Mutant Advanced NSCLC
Acronym: CURCUMIN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Davis Institute (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Victor Cohen, MD,CM, FRCPC, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: JGH-14-149
Record Dates: First submitted 2014-12-01; First posted 2014-12-22 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: curcumin; lung cancer; TKI
MeSH Terms: conditions — Lung Neoplasms | interventions — Curcumin; Gefitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CurcuVIVA™ (NPN 80027414) at a single dose of 80 mg PO daily without any dose escalation to be taken in conjunction with an EGFR-TKI therapy.
  CurcuVIVA™ is given in capsule forms. Unit strength of CurcuVIVA™ is equal to Turmeric Extract 25:1 348 mg (containing 80mg Longvida® Optimized Curcumin)
  Tyrosine Kinase Inhibitors:
  1. Gefitinib is a targeted therapy, given in a capsule form once daily. The daily dose is 250 mg .
  2. Erlotinib is a targeted therapy, given in a capsule form once daily. The daily dose is 150 mg .
  Study intervention is 8 weeks, following which the patients will continue taking their EGFR-TKI without curcumin until progression. The side effects of curcumin will be followed for another 8 weeks from the date of stopping curcumin.
  Interventions: Dietary Supplement: CurcuVIVA™; Drug: Tyrosine Kinase Inhibitor gefitinib (Iressa); Drug: Tyrosine Kinase Inhibitor erlotinib (Tarceva)

INTERVENTIONS:
Dietary Supplement: CurcuVIVA™ — 80 mg PO daily for 8 weeks with an option to reduce the dose based on individual tolerability
  Other Names: Curcumin
Drug: Tyrosine Kinase Inhibitor gefitinib (Iressa) — 250 mg PO daily until progression
  Other Names: gefitinib (Iressa)
Drug: Tyrosine Kinase Inhibitor erlotinib (Tarceva) — 150 mg PO daily until progression
  Other Names: erlotinib (Tarceva)

SUMMARY:
The purpose of this study is is to assess the safety and tolerability of curcumin in combination with EGFR-TKIs in selected patients with advanced non-resectable mutant EGFR NSCLC.

DETAILED DESCRIPTION:
This is a phase 1 open prospective cohort study to assess the safety and feasibility of using curcumin in conjunction with an EGFR-TKI in patients with advanced NSCLC. The investigators will use an enhanced bioavailable formulation of curcumin (CURCUViva TM at 80 mg/ 1 capsule per day) approved and licensed by Health Canada (NPN 80027414) that has been shown to have 2-3 times higher curcumin concentration in the blood as compared to previous clinical trials. As primary objective, the investigators will recruit 20 patients for a duration of 8 weeks to monitor adverse effects according to the the National Cancer Institute Common Terminology Criteria.Exploratory objectives would include assessing changes in health-related quality of life using the standardized FACT-L questionnaire and evaluating anti-inflammatory properties of curcumin by measuring CRP. If tolerable safety data is obtained, an expanded phase II trial will be designed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or patients on treatment for histologically confirmed advanced EGFR-mutant NSCLC defined as unresectable stage 3A, stage 3B or stage 4.
* The EGFR mutation analysis must be performed prior to enrolment into the trial (i.e., before a patient is consented). Any EGFR mutation-positive result must be documented and the analysis for the mutation will be performed using the JGH local testing methodology.
* Receiving concurrent EGFR-TKI therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0-3

Exclusion Criteria:

* Symptomatic brain metastases.
* Patients who are receiving any other investigational agents.
* Patients using other non-vitamin or mineral regular natural health product, which includes Chinese Herbs.
* Incapacity to understand and sign a written informed consent document in English/French.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
feasibility assessed by: Willingness of patients to participate= Number of enrolled/Number of approached patients, | 8 weeks
  Feasibility will determine whether the use of curcumin is appropriate for further testing; and will be assessed by:
  Willingness of patients to participate= Number of enrolled/Number of approached patients,
feasibility assessed by follow-up rate= number of actual study visits/ total number of study visits | 8 weeks
  will by assessed by follow-up rate= number of actual study visits/ total number of study visits
feasibility Adherence/Compliance rate= Number of taken capsules/Total number of capsules | 8 weeks
  Adherence/Compliance rate= Number of taken capsules/Total number of capsules
feasibility Questionnaires completion rate= Number of completed questionnaires/Total number of questionnaires | 8 weeks
  Questionnaires completion rate= Number of completed questionnaires/Total number of questionnaires
safety number of side effects | 16 weeks
  Safety will be assessed by number of side effects

SECONDARY OUTCOMES:
To evaluate and compare the changes in health-related quality of life before and after | 8 weeks
  Patients' quality of life on curcumin treatment will be assessed by the FACT-L at the baseline, 4 weeks,8 weeks on concurrent curcumin and TKI and 8 weeks post-study. Clinically important difference in the score is considered 2 points.
To evaluate anti-inflammatory properties of Curcumin (assessed by measuring C-reactive protein) | 8 weeks
  anti-inflammatory effects of curcumin will be assessed by measuring C-reactive protein tests will be performed at baseline, 2, 4, 8 and 16 weeks into study.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Cohen, MD, Principal Investigator — Lady Davis Institute
Locations (1):
- Peter Brojge Lung Cancer Center, Jewish General Hospital, Montreal, Quebec, Canada